CLINICAL TRIAL: NCT01203358
Title: Efficacy and Safety of Exosurf Neonatal and Survanta for the Treatment of Respiratory Distress Syndrome
Brief Title: Exosurf Neonatal and Survanta for Treatment of Respiratory Distress Syndrome
Acronym: Surfactant 1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Responsible Party: Jeffrey D. Horbar/ Lead Principal Investigator, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0003; U01HD019897 (NIH); U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD021397 (NIH); U10HD021415 (NIH); U10HD027856 (NIH); U10HD027853 (NIH); U10HD027871 (NIH); U10HD027851 (NIH); U10HD027880 (NIH); U10HD027881 (NIH)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Bronchopulmonary Dysplasia
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Respiratory distress syndrome; Surfactant
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome | interventions — dipalmitoylphosphatidylcholine, hexadecanol, tyloxapol drug combination; beractant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surfactant 1 (Active Comparator): Exosurf Neonatal (Burroughs Wellcome Co.)
  Interventions: Drug: Exosurf
- Surfactant 2 (Active Comparator): Survanta (Ross Laboratories)
  Interventions: Drug: Survanta

INTERVENTIONS:
Drug: Exosurf — Infants received up to four intratracheal doses of the surfactant.
  Other Names: Exosurf Neonatal (Burroughs Wellcome Co.)
  Arms: Surfactant 1
Drug: Survanta — Infants received up to four intratracheal doses of the surfactant.
  Other Names: Survanta (Ross Laboratories)
  Arms: Surfactant 2

SUMMARY:
The purpose of this study is to compare the efficacy of two surfactants, Exosurf Neonatal (Burroughs Wellcome Co.) and Survanta (Ross Laboratories), for the treatment of neonatal respiratory distress syndrome.

DETAILED DESCRIPTION:
The NICHD Neonatal Research Network conducted a randomized trial at 11 centers comparing the efficacy of two surfactants -- Exosurf Neonatal (Burroughs Wellcome Co.) and Survanta (Ross Laboratories) -- for the treatment of neonatal respiratory distress syndrome. Newborn infants with birth weights of 501-1500g with respiratory distress syndrome who were receiving assisted ventilation with 30% oxygen or more within 6 hours of birth were enrolled between January 1991 and January 1992. Infants were randomly assigned to receive up to four intratracheal doses of either Exosurf Neonatal or Survanta.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants weighing 501 to 1500 gm with respiratory distress syndrome were receiving assisted ventilation with 30% oxygen or more

Exclusion Criteria:

* Less than 6 hours of age

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 617 (Actual)
Dates: Start 1991-01; Primary Completion 1992-01 (Actual); Study Completion 1992-01 (Actual)

PRIMARY OUTCOMES:
Death or bronchopulmonary dysplasia | 28 days of life

SECONDARY OUTCOMES:
Average fraction of inspired oxygen (FIO2) | 72 hours after treatment
Mean airway pressure (MAP) | 72 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D. Horbar, MD, Study Director — University of Vermont; Elizabeth C. Wright, PhD, Principal Investigator — George Washington University; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Charles R. Bauer, MD, Principal Investigator — University of Miami; Jon E. Tyson, MD MPH, Principal Investigator — University of Texas; James A. Lemons, MD, Principal Investigator — Indiana University; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Barbara J. Stoll, MD, Principal Investigator — Emory University; David K. Stevenson, MD, Principal Investigator — Stanford University; LuAnn Papile, MD, Principal Investigator — University of New Mexico
Locations (13):
- United States (13):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Result] Horbar JD, Wright LL, Soll RF, Wright EC, Fanaroff AA, Korones SB, Shankaran S, Oh W, Fletcher BD, Bauer CR, et al. A multicenter randomized trial comparing two surfactants for the treatment of neonatal respiratory distress syndrome. National Institute of Child Health and Human Development Neonatal Research Network. J Pediatr. 1993 Nov;123(5):757-66. doi: 10.1016/s0022-3476(05)80856-x. PMID 8229487
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/